CLINICAL TRIAL: NCT04444310
Title: Antibody Responses in Asymptomatic Close Contacts of COVID-19 Patients and Their Implications
Brief Title: Antibody Responses in Contacts of COVID-19 Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Aliae AR Mohamed Hussein, Professor of Pulmonology, Assiut University
Other Study IDs: Assiut13
Record Dates: First submitted 2020-06-19; First posted 2020-06-23 (Actual); Last update posted 2020-06-23 (Actual); Status verified 2020-06

CONDITIONS: COVID-19
Keywords: COVID-19; antibodies; IgG; IgM; SARs-CoV-2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 14 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After several cases of pneumonia with an unfamiliar etiology were observed at the end of 2019, the National Health Commission of China released more details about the epidemic in early 2020. The pathogen was identified as a novel coronavirus and named severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), as it has a phylogenetic similarity to SARS-CoV. Since then, SARS-CoV-2 has spread rapidly and the resulting coronavirus disease 2019 (COVID-19) has been declared a public health emergency of international concern (PHEIC) by the World Health Organization (WHO).

SARS-CoV-2 is highly contagious, and there has not yet been any vaccine or effective treatment that has received approval. So, the best solution for controlling the pandemic will be the simultaneous application of preventive methods, sensitive diagnostic approaches, and using current available drugs, while still developing novel treatments.

Coronaviruses are enveloped, non-segmented, single positive-stranded RNA viruses with round or oval particles and a diameter of 50-200 nm. Coronavirus subfamily is divided into four genera: α, β, γ and δ according to serotype and genomic characteristics.

DETAILED DESCRIPTION:
The SARS-CoV-2 belongs to the genus β which has been confirmed to be highly infectious by research. (https://www.who.int/emergencies/ diseases/novel-coronavirus-2019/situation-reports).

The four major structural proteins of coronavirus are the spike surface glycoprotein (S), small envelope protein (E), matrix protein (M), and nucleocapsid protein (N). The spike protein (S) of coronavirus is a type I transmembrane glycoprotein and mediates the entrance to human respiratory epithelial cells by interacting with cell surface receptor angiotensin-converting enzyme 2 (ACE2) , the S protein contains distinct functional domains near the amino (S1) and carboxy (S2) termini, the peripheral S1 portion can independently bind cellular receptors while the integral membrane S2 portion is required to mediate fusion of viral and cellular membranes . The nucleocapsid protein (N) forms complexes with genomic RNA, interacts with the viral membrane protein during virion assembly and plays a critical role in enhancing the efficiency of virus transcription and assembly .

The diagnosis of COVID-19 is dependent mainly on clinical characteristics, CT imaging and a few laboratory tests. Although some symptoms and laboratory parameters have indicative values in confirmed patients, they are not unique to SARSCoV-2 infection. The most used and reliable test for diagnosis of COVID-19 has been the RT-PCR test performed using nasopharyngeal swabs. A variety of RNA gene targets are used by different manufacturers, with most tests targeting 1 or more of the envelope (env), nucleocapsid (N), spike (S), RNA-dependent RNA polymerase (RdRp), and ORF1 genes .

Spread of the COVID-19 global pandemic highlights the urgent need to develop effective treatments or vaccines against SARS-CoV-2 infection. The identification of novel antibodies to neutralize the virus is one of the approaches to fight COVID-19 . In particular, detect an antibody against the SARS-CoV-2 spike protein by building on knowledge about the existing structure of SARS-CoV-2 and learnings from previous SARS antibody generations. Potent neutralizing antibodies often target the receptor interaction site in S1, disabling receptor interactions. The so-called spike protein of 2019-nCoV is used by the virus to dock to human cells. By targeting the protein, to prevent the infection.

COVID-19 patients developed SARS-CoV-2-specific NAbs at the convalescent phase of infection (SARS-CoV-2 NAbs were unable to cross-reactive with SARS-CoV virus). SARS-CoV -2 specific NAbs reached their peak in patients from day 10-15 after the onset of the disease and remained stable thereafter in the patients. Antibodies targeting on different domains of S protein, including S1, RBD, and S2, may all contribute to the neutralization.

Neutralizing antibodies (NAbs) play important roles in virus clearance and have been considered as a key immune product for protection or treatment against viral diseases. Virus-specific NAbs, induced through either infection or vaccination, can block viral infection . NAbs confer immunity by deactivate viruses by block access to receptors used by the virus to enter host cells and bind to viral capsid and block uncoating of the viral genome .

The level of NAbs has been used as a gold standard to evaluate the efficacy of vaccines against smallpox, polio and influenza viruses . Passive antibody therapy, such as plasma fusion, was successfully used to treat infectious viral diseases, including SARS-CoV virus, influenza viruses, and Ebola virus. The efficacy of passive antibody therapy was associated with the concentration of NAbs in plasma or antibodies of recovered donors. As the global pandemic of COVID-19 proceeds, transfusion of convalescent plasma or serum from recovered patients was also considered as a promising therapy for prophylaxis of infection or treatment of disease. highly variable levels of NAbs in the patients of COVID-19 indicated that convalescent plasma and serum from recovered donors should be titrated before use in passive antibody therapy, an easy task that can be performed using the PsV neutralization assay. The titers of NAbs were variable in different patients. Elderly patients (60-80 ys) were more likely to induce higher titers of NAbs than younger patients. A moderate positive correlation was also observed between age and Nab titers confirming the important role of age in the generation of Nabs. The correlation of NAbs titers with age, lymphocyte counts, and blood CRP levels suggested that the interplay between virus and host immune response.

ELIGIBILITY:
Inclusion Criteria:

* close contacts of confirmed COVID-19 patients, apparently healthy

Exclusion Criteria:

* symptomatic close contacts, any close contacts with malignant tumor, stroke, cardiac, respiratory, Gastrointestinal, and renal diseases or any organ dysfunction.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: asymptomatic close contacts of confirmed COVID-19 patients, not complaining
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-06-15 (Actual); Primary Completion 2020-06-18 (Actual); Study Completion 2020-09-30 (Estimated)

PRIMARY OUTCOMES:
Measure level of Abs in asymptomatic close contacts of COVID 19 patients. | one day
  serum level of antiSARS-CoV-2 IgG, IgM

CONTACTS AND LOCATIONS:
Locations (1):
- AssiutU, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided